CLINICAL TRIAL: NCT00891371
Title: A Phase II-III, Multicentre, Prospective, Exploratory, Open Label Study to Assess the Efficacy and Safety of Lanreotide Autogel 120mg in the Symptomatic Treatment of Patients With Refractory Diarrhea
Brief Title: Lanreotide Autogel in the Symptomatic Treatment of Refractory Diarrhea
Acronym: MEDARD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-48-52030-223; 2009-009356-20 (EudraCT Number)
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Diarrhea
Keywords: symptomatic treatment of patients with refractory diarrhea
MeSH Terms: conditions — Diarrhea | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lanreotide (Autogel formulation) Autogel 120mg (Experimental): lanreotide (Autogel formulation) Autogel 120mg
  Interventions: Drug: lanreotide (Autogel formulation)

INTERVENTIONS:
Drug: lanreotide (Autogel formulation) — Autogel 120mg

SUMMARY:
The purpose of this study, is to assess the effect of lanreotide Autogel 120mg on stool frequency in subjects with refractory diarrhea at day 28 (mean of last 7 days) compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Male/female with refractory diarrhea for at least 1 month, after normal extended work-up to exclude causes of diarrhea, not or not enough responding to standard anti-diuretics as evaluated by the investigator
* Patient mentally fit for completing a diary

Exclusion Criteria:

* Has already received a treatment with somatostatin analogues for the treatment of refractory diarrhea
* Had a weight of stool < 600g in a 72hrs stool collection
* Has received a treatment with laxatives within the last week before study entry
* Suffers from IBS with alternating bowel habits and predominant constipation, suffers from infectious and/or inflammatory gastro-enteritis (colitis ulcerosa, crohn's disease and macroscopic colitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (11):
- Belgium (11):
  - OLVZ Aalst, Aalst
  - ZNA Antwerpen, Antwerp
  - AZ Sint Lucas Brugge, Bruges
  - UZ Antwerpen #2, Edegem
  - ZOL, Genk
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHC Cliniques Saint Joseph, Liège
  - CHU A. Vesale, Montigny-le-Tilleul
  - AZ Sint-Augustinus, Wilrijk

REFERENCES:
- [Derived] Bisschops R, De Ruyter V, Demolin G, Baert D, Moreels T, Pattyn P, Verhelst H, Lepoutre L, Arts J, Caenepeel P, Ooghe P, Codden T, Maisonobe P, Petrens E, Tack J. Lanreotide Autogel in the Treatment of Idiopathic Refractory Diarrhea: Results of an Exploratory, Controlled, Before and After, Open-label, Multicenter, Prospective Clinical Trial. Clin Ther. 2016 Aug;38(8):1902-1911.e2. doi: 10.1016/j.clinthera.2016.06.012. Epub 2016 Aug 8. PMID 27423779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicentered study performed at 18 investigational sites in Belgium of which 11 recruited patients.
Groups:
- Lanreotide Autogel 120 mg: Lanreotide Autogel 120 mg one subcutaneous injection on Day 1 and Day 28.
Period: Pre-assignment
Arm/Group | Lanreotide Autogel 120 mg
Started | 42
Completed | 36
Not Completed | 6
Not completed — Inclusion/exclusion | 5
Not completed — Consent withdrawal | 1
Period: Treatment
Arm/Group | Lanreotide Autogel 120 mg
Started | 36
Completed | 27
Not Completed | 9
Not completed — Lack of Efficacy | 5
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The Safety population was defined as all subjects who received at least one injection of the study medication.
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (16.4)
Age, Customized [Number; unit: participants]
  <30 years | 2
  >=30 to <65 years | 22
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 12
Race [Caucasian / White] [Number; unit: Participants] | 36
Quality Of Life (QOL) - Scales [Mean (Standard Deviation); unit: units on a scale] — SF36 QOL includes 1 multi-item scale measuring each of 8 health concepts. These scores are summed to produce raw scale scores for each health concept which are transformed to a 0-100 scale. There is in addition a single-item measure of Health Transition
  IBS-QOL is a self-report QOL measure specific to IBS that can be used to assess impact of IBS and its treatment. This consists of 34 items,each with a 5 point response scale.Individual responses to 34 items are summed and averaged for a total score and transformed to a 0-100 scale with higher scores indicating better IBS specific QOL
  units on a scale
    SF36 QOL: Physical Functioning | 60.5 (29.1)
    SF36 QOL: Role Physical | 39.6 (30.9)
    SF36 QOL: Role Emotional | 52.8 (38.7)
    SF36 QOL: Vitality | 38.8 (24.1)
    SF36 QOL: Mental Health | 47.6 (23.1)
    SF36 QOL: Social Functioning | 41.1 (31.2)
    SF36 QOL: Bodily Pain | 48.7 (30.4)
    SF36 QOL: General Health | 43.9 (22.8)
    IBS QOL: Total Score | 47.4 (18.5)
Score of Stool Consistency (Bristol Stool Form Scale) [Median (Full Range); unit: units on a scale] — Each patient scored his/her stool on the Bristol Stool Form Scale: Type 1 - Separate hard lumps, like nuts (hard to pass); Type 2 - Sausage-shaped but lumpy; Type 3 - Like a sausage but with cracks on its surface; Type 4 - Like a sausage or snake, smooth and soft; Type 5 - Soft blobs with clear-cut edges (passed easily); Type 6 - Fluffy pieces with ragged edges, a mushy stool; Type 7 - Water no solid pieces, Entirely liquid
  units on a scale | 6.0 [5 to 7]
Mean Number of Stools [Mean (Standard Deviation); unit: Number of Stools] | 5.5 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Having Minimum Reduction of 50% or Normalization (≤3 Stools/24hours) in the Mean Number of Stools (Mean of Last 7 Days)
Time Frame: Day 28
Population: Intention to Treat (ITT) Population [All treated subjects with at least 3 Days of available primary efficacy variable data for both Baseline and post Baseline periods]
Measure: Number; unit: Percentage of patients
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 36
Percentage of patients
  Reduction of at least 50% or normalization - Yes | 44.4
  Reduction of at least 50% or normalization - No | 55.6

2. Secondary Outcome: Change in QOL-Quality of Life {Assess Using Short Form (SF-36) and Irritable Bowel Syndrome (IBS)-QOL} Compared to Baseline
Description: SF36 QOL includes 1 multi-item scale measuring each of 8 health concepts. These scores are summed to produce raw scale scores for each health concept which are transformed to a 0-100 scale. The lower the score the more disability. The higher the score the less disability. There is in addition a single-item measure of Health Transition
  IBS-QOL is a self-report QOL measure specific to IBS that can be used to assess impact of IBS and its treatment. This consists of 34 items,each with a 5 point response scale.Individual responses to 34 items are summed and averaged for a total score and transformed to a 0-100 scale with higher scores indicating better IBS specific QOL
Time Frame: Baseline (Day 1), Day 21, Day 28, Day 49 and Day 56
Population: ITT Population, Analysis based on number (n) of patients with a valid value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 36
units on a scale
  SF36 QOL: Physical Functioning (D21), n=33 | -1.3 (20.5)
  SF36 QOL: Physical Functioning (D28), n=34 | 2.4 (19.6)
  SF36 QOL: Physical Functioning (D49), n=26 | 2.9 (18.9)
  SF36 QOL: Physical Functioning (D56), n=35 | 1.1 (23.3)
  SF36 QOL: Role Physical (D21), n=33 | 4.5 (19.6)
  SF36 QOL: Role Physical (D28), n=34 | 12.9 (21.8)
  SF36 QOL: Role Physical (D49), n=26 | 6.3 (28.3)
  SF36 QOL: Role Physical (D56), n=35 | 11.8 (23.5)
  SF36 QOL: Role Emotional (D21), n=33 | -0.3 (34.8)
  SF36 QOL: Role Emotional (D28), n=34 | 3.4 (40.7)
  SF36 QOL: Role Emotional (D49), n=25 | 7.0 (35.2)
  SF36 QOL: Role Emotional (D56), n=35 | 5.0 (39.6)
  SF36 QOL: Vitality (D21), n=32 | 3.1 (22.1)
  SF36 QOL: Vitality (D28), n=33 | 5.9 (22.2)
  SF36 QOL: Vitality (D49), n=24 | 2.1 (24.6)
  SF36 QOL: Vitality (D56), n=34 | 7.2 (23.9)
  SF36 QOL: Mental Health (D21), n=32 | 5.8 (27.9)
  SF36 QOL: Mental Health (D28), n=33 | 8.3 (28.2)
  SF36 QOL: Mental Health (D49), n=24 | 8.3 (27.1)
  SF36 QOL: Mental Health (D56), n=34 | 10.1 (27.7)
  SF36 QOL: Social Functioning (D21), n=31 | 9.3 (27.8)
  SF36 QOL: Social Functioning (D28), n=33 | 16.7 (29.8)
  SF36 QOL: Social Functioning (D49), n=24 | 19.3 (34.8)
  SF36 QOL: Social Functioning (D56), n=33 | 14.0 (31.5)
  SF36 QOL: Bodily Pain (D21), n=33 | -4.6 (31.5)
  SF36 QOL: Bodily Pain (D28), n=34 | 8.3 (28.6)
  SF36 QOL: Bodily Pain (D49), n=26 | 8.8 (29.2)
  SF36 QOL: Bodily Pain (D56), n=35 | 5.3 (30.7)
  SF36 QOL: General Health (D21), n=33 | -2.8 (16.0)
  SF36 QOL: General Health (D28), n=33 | 2.8 (16.8)
  SF36 QOL: General Health (D49), n=26 | 4.1 (19.1)
  SF36 QOL: General Health (D56), n=34 | 3.7 (19.9)
  IBS QOL: Total Score (D21), n=27 | 9.9 (21.5)
  IBS QOL: Total Score (D28), n=26 | 13.9 (22.0)
  IBS QOL: Total Score (D49), n=22 | 16.8 (22.5)
  IBS QOL: Total Score (D56), n=29 | 16.3 (22.5)

3. Secondary Outcome: Change in Median Score of Stool Consistency (Bristol Stool Form Scale) Compared to Baseline
Description: Each patient scored his/her stool on the Bristol Stool Form Scale: Type 1 - Separate hard lumps, like nuts (hard to pass); Type 2 - Sausage-shaped but lumpy; Type 3 - Like a sausage but with cracks on its surface; Type 4 - Like a sausage or snake, smooth and soft; Type 5 - Soft blobs with clear-cut edges (passed easily); Type 6 - Fluffy pieces with ragged edges, a mushy stool; Type 7 - Water no solid pieces, Entirely liquid
Time Frame: Baseline (day 1), day 28 and day 56
Population: ITT Population; Missing number of subjects = 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 35
units on a scale
  Change from Baseline to Day 28 | 0.0 [-3 to 1]
  Change from Baseline to Day 56 | -0.5 [-4 to 1]

4. Secondary Outcome: Percent Change in Mean Number of Stools Compared to Baseline
Time Frame: Baseline (Day 1), Day 28 and Day 56
Population: ITT Population; Missing number of subjects = 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 35
Percent change
  Change from Baseline to Day 28 | -25.9 (36.7)
  Change from Baseline to Day 56 | -30.7 (38.0)

5. Secondary Outcome: Change From Baseline in Relative Frequency of Normalization (≤3 Stools) in Subjects
Description: Normalization of stool frequency in subjects with refractory diarrhoea at Day 28 and Day 56 (mean of last 7 days) compared to Baseline.
Time Frame: Baseline (Day 1), Day 28 and Day 56
Population: ITT Population; Missing number of subjects = 1
Measure: Mean (Standard Deviation); unit: Percentage of days per Week
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 35
Percentage of days per Week
  Change from Baseline to Day 28 | 27.5 (34.7)
  Change from Baseline to Day 56 | 33.0 (34.3)

6. Secondary Outcome: Percentage of Patients Having Minimum Reduction of At Least 50% or Normalization of the Mean Number of Stools
Time Frame: Day 56
Population: ITT Population; Missing number of subjects: 1
Measure: Number; unit: Percentage of participants
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 35
Percentage of participants
  Reduction of at least 50% or normalization - Yes | 54.3
  Reduction of at least 50% or normalization - No | 45.7

ADVERSE EVENTS:
Time Frame: Up to Day 56 (± 2)
Description: Treatment Emergent Adverse Events (TEAE)
Arm/Group | Lanreotide Autogel 120 mg
Serious Adverse Events (participants affected / at risk) | 5/36
Other Adverse Events (participants affected / at risk) | 30/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel 120 mg (N=36)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Steatorrhoea (Gastrointestinal disorders) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel 120 mg (N=36)
Abdominal pain (Gastrointestinal disorders) | 9 (10)
Constipation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Steatorrhoea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 4 (4)
Influenza like illness (General disorders) | 2 (3)
Injection site nodule (General disorders) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (5)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes